CLINICAL TRIAL: NCT01454037
Title: Immune Profiles and Circulating Tumor Cell Status Following Prostate Cryotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201107059RB
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer; Immune Profile; Circulating Cancer Cells; Clinical Corelation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Prostate cryoablation: Subjects receiving cryotherapy for prostate cancer
  Interventions: Procedure: Prostate cryotherapy
- Radical prostatectomy: Subjects receiving radical prostatectomy
  Interventions: Procedure: Radical prostatectomy
- Radiation: Subjects receiving radiation for prostate cancer
  Interventions: Procedure: Radiation

INTERVENTIONS:
Procedure: Prostate cryotherapy — cryoablate the prostate
  Groups: Prostate cryoablation
Procedure: Radical prostatectomy — Remove prostate
  Groups: Radical prostatectomy
Procedure: Radiation — Radiate prostate
  Groups: Radiation

SUMMARY:
The change of immune profiles and existence of circulating tumor cells following prostate cryotherapy may be correlated with the clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age>20 years
* Histopathology-proven prostate adenocarcinoma
* Non-metastatic localized disease
* Subjects have chosen their curative, definitive treatments for prostate cancer prior to enrolling for the study
* Subjects are willing to sign the informed consent and agree to comply with the study procedures

Exclusion Criteria:

* Chronic use (> 2 weeks) of > 10 mg/day of prednisone or prednisolone within 2 months of the screening (topical or inhalational corticosteroids are permitted)
* Concurrent use of immunosuppressive therapy, including: cyclosporine, antithymocyte globulin, or tacrolimus within 3 months of study entry
* Other conditions the investigators think may affect subjects' compliance

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taiwanese organ-confined or locally advanced prostate cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Cancer recurrence | 3, 6, 12, 24 months after treatments
  Includes:
  1. Biochemical (PSA) recurrence according to the ASTRO or Phoenix criteria for patients undergoing cryotherapy (Cryo) or radiotherapy (RT)
  2. Prostate biopsy positivity
  3. Radiographic evidence of recurrence (CT/MRI, Bone scan, radiographs, etc.) Time to recurrence defined by the either of the above 3 outcome parameters

SECONDARY OUTCOMES:
Quality of life | 3, 6, 12, 24months after treatments
  according to the QLQ C30 and PR25 questionnaire interview

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan